CLINICAL TRIAL: NCT07155447
Title: Perioperative Nutrition Optimization for Reducing Complications After Surgical Fracture Fixation
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 33444
Record Dates: First submitted 2025-02-23; First posted 2025-09-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Lower Extremity Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients randomized to CEAA (Experimental): Patients with lower extremity fractures indicated for operative fracture fixation at six tertiary trauma centers
  Interventions: Dietary Supplement: CEAA supplementation
- patients randomized to placebo (Placebo Comparator): Patients with with lower extremity fractures indicated for operative fracture fixation at six tertiary trauma centers
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CEAA supplementation — (including calcium beta-hydroxy-beta- methylbutyrate monohydrate, L-Arginine, L-Glutamine and Ciltruline) Supplementation will be started within 72 hours of presentation and continued for a period of 28 days.
  Arms: Patients randomized to CEAA
Other: Placebo — a neutral powder containing the non- essential amino acid Alanine which will be indistinguishable from the CEAA supplement powder in in regards to packaging and supplement appearance.
  Arms: patients randomized to placebo

SUMMARY:
The objective of this multi-center, prospective, placebo-controlled, randomized study is to compare oral conditionally essential amino acid (CEAA) supplementation for decreasing the key postoperative complications of fracture-related infection, fracture nonunion, and skeletal muscle wasting with a placebo control (PC) after lower extremity fracture fixation. Investigators hypothesize that perioperative oral supplementation with an investigational CEAA supplement (ICS) will reduce postoperative fracture-related infections, fracture nonunion rates, and skeletal muscle wasting in patients with traumatic lower extremity fractures. This is supported by strong pilot data. Conducting a randomized controlled trial at five civilian tertiary referral centers and one military treatment facility will further study the potential benefits of oral CEAA supplementation for preventing the stated key postoperative complications in patients following high energy lower extremity orthopedic trauma. This low cost, low risk intervention has demonstrated potential to expedite Warfighter return to duty as well as potentially reducing delayed limb amputations and mortality in severely injured patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18-55 years
2. Open or closed fracture of the lower extremity including femur, tibia and/or fibula, calcaneus, talus, Lisfranc joint (OTA/AO 31, 32, 33, 41, 42, 43, 44, 4F, 81, 82, 83, 85)
3. Ability to begin supplementation within 72 hours of injury

Exclusion Criteria:

1. BMI <18.5 kg/m 2 (underweight) or BMI > 45 kg/m 2 (severe obesity) to exclude patients with severely increased baseline risk of adverse outcome due to preoperative poor nutrition
2. Non-ambulatory prior to injury
3. Currently pregnant
4. Medical contraindication to CEAA supplementation (e.g., phenylketonuria)
5. Inability to provide informed consent due to intellectual disability
6. Protected populations (e.g., prisoners)
7. Inability to follow up (e.g., homeless at time of surgery, home address out of state of treating facility)
8. Documented dementia, mild or moderate traumatic brain injury
9. Inability to consume supplement or placebo due to head or neck trauma
10. Low-energy fragility fracture (i.e. ground level falls)
11. Pathologic fracture (i.e. fracture through site of compromised bone due to infection, neoplasm, documented osteoporosis, metabolic bone disease from conditions such as end stage renal disease, osteomalacia, hypophosphatemic rickets, renal osteodystrophy, osteofibrous dysplasia)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare clinical benefit of oral supplementation with CEAA versus a placebo for reducing fracture-related infection after lower extremity fracture fixation. | 12 months
  Investigators will record the number of participants with fracture-related infection for 12 months following lower extremity fracture fixation. The measurement will be based on Metsemakers consensus definition (Metsemakers et al. (2018). We will enroll 1,000 participants and anticipate 15% loss to attrition (426 in each arm).
  Using the observed fracture-related infection rates of 16.5% and 10% from a previous study, 426 participants would be needed for each group to detect a significant difference with 80% power and alpha value of 0.05 based upon Pearson Chi-Square test and pooled standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Hendrickson, Principal Investigator — University of Minnesota